CLINICAL TRIAL: NCT03279341
Title: An Open-label, Randomised, Crossover, Reader Blinded, Study to Compare the Effect of Polyethylene Glycol 3350, Bisacodyl and Prucalopride on Colonic Motility Assessed With Intraluminal Colonic Manometry in Healthy Subjects
Brief Title: Effect of PEG, Bisacodyl and Prucalopride on Colonic Motility in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Maura Corsetti, Associate Professor of Gastroenterology, University Hospital, Gasthuisberg
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: S54750
Record Dates: First submitted 2017-08-22; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Chronic Constipation
Keywords: laxatives; constipation
MeSH Terms: conditions — Constipation | interventions — Polyethylene Glycols; Bisacodyl; prucalopride

STUDY DESIGN:
Intervention Model Description: open-label, randomized, reader-blinded, 3-period cross-over study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- polyethylene glycol, osmotic laxitive (Active Comparator): 13.8g polyethylene glycol 3350 with sodium bicarbonate, sodium chloride, and potassium chloride, mixed with 125mL of water administered twice orally as a solution
  Interventions: Drug: polyethylene glycol
- bisacodyl, stimulant laxative (Active Comparator): 10 mg bisacodyl once daily oral administration with 125mL of water
  Interventions: Drug: Bisacodyl
- prucalopride, prokinetic (Active Comparator): 2mg prucalopride, film-coated tablets (prucalopride succinate eq. 2mg), once daily oral administration with 125mL of water
  Interventions: Drug: Prucalopride

INTERVENTIONS:
Drug: polyethylene glycol — osmotic laxative
  Other Names: macrogol; PEG
  Arms: polyethylene glycol, osmotic laxitive
Drug: Bisacodyl — stimulant laxative
  Other Names: Dulcolax
  Arms: bisacodyl, stimulant laxative
Drug: Prucalopride — prokinetic
  Other Names: Resolor
  Arms: prucalopride, prokinetic

SUMMARY:
This study aim was to evaluate the effect of pharmacological treatments normally used to treat functional constipation and in particular PEG, bisacodyl and prucalopride on colonic motility as assessed by high-resolution manometry.

DETAILED DESCRIPTION:
Rationale: Several treatments with different modes of action are currently available for chronic constipation. This study will investigate the effect of these different modes of actions of PEG 3350 + electrolytes, bysacodyl and prucalopride and on colonic motility parameters (e.g. HAPC).

Objectives:Primary: to compare and determine the effects of PEG, bisacodyl and prucalopride on the number of colonic high amplitude propagated contractions (HAPCs) during a 12-hour intraluminal manometry in healthy subjects. Secondary: to evaluate the association between motility parameters and number and consistency of bowel movements in healthy subjects.

Investigational product, dose, and mode of administration: Regimen A: 13.8g polyethylene glycol 3350 with sodium bicarbonate, sodium chloride, and potassium chloride, mixed with 125mL of water administered twice orally as a solution. Regimen B: 10 mg bisacodyl once daily oral administration with 125mL of water. Regimen C: 2mg prucalopride, film-coated tablets (prucalopride succinate eq. 2mg), once daily oral administration with 125mL of water.

Methodology: This is an open-label, randomized, reader-blinded, 3-period cross-over study investigating the effects of PEG 3350 + electrolytes, bisacodyl and prucalopride on colon motility with intraluminal manometry. On day 1 of each Treatment Period, a manometry catheter will be placed in the colon under conscious sedation and the colonic pressure will be continuously measured through 12 hours after administration of each of the investigational products (Regimen A, B or C).

Inclusion criteria: healthy male and non-pregnant, non-breastfeeding female participants, aged 18-65 years old at the time of consent. Exclusion criteria: use of medications within 48 h of dose initiation; structural or metabolic diseases that affect the gastrointestinal system and functional gastrointestinal disorders; previous abdominal surgery other than appendectomy, cholecystectomy, hysterectomy, or hernia repair; known illnesses such as diabetes, cardiovascular or lung disease; use of agents that influence bowel habit, i.e. anticholinergics (not including antihistamines with anticholinergic properties), spasmolytics and prokinetics in the 7 days before the study.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and non-pregnant, non-breastfeeding female participants, aged 18-65 years old at the time of consent

Exclusion Criteria:

* use of medications within 48 h of dose initiation; structural or metabolic diseases that affect the gastrointestinal system and functional gastrointestinal disorders; previous abdominal surgery other than appendectomy, cholecystectomy, hysterectomy, or hernia repair; known illnesses such as diabetes, cardiovascular or lung disease; use of agents that influence bowel habit, i.e. anticholinergics (not including antihistamines with anticholinergic properties), spasmolytics and prokinetics in the 7 days before the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-12-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
colonic motor patterns during PEG, bisacodyl and prucalopride in healthy subjects. | during a 12-hour intraluminal manometry
  number of colonic high amplitude propagated contractions (HAPCs)

SECONDARY OUTCOMES:
association between motility parameters and number and consistency of bowel movements in healthy subjects | during a 12-hour intraluminal manometry
  number of colonic motor patterns and number of bowel movements and stool consistency assessed by Bristol Stool Chart

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD. PhD, Principal Investigator — KU Leuven
Locations (1):
- TARGID, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No